CLINICAL TRIAL: NCT07296419
Title: Dual System Study: Transvaginal Fetal Pulse Oximetry Measurement Systems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raydiant Oximetry, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP2555
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Fetal Hypoxia; Fetal Acidemia
MeSH Terms: conditions — Fetal Hypoxia

STUDY DESIGN:
Intervention Model Description: The Raydiant Oximetry Data Collection System (DCS) generates waveforms representing fetal SpO2. In this study, the objective is to compare the waveforms generated by the DCS to the Nellcor N-400 actual fetal SpO2 values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Dual Sensor Recipients (Experimental): Women in labor who consent to participation are monitored using two sterile fetal sensors and two separate data collection systems.
  Interventions: Device: Fetal Pulse Oximetery

INTERVENTIONS:
Device: Fetal Pulse Oximetery — Two fetal pulse oximeter sensors are connected to two separate systems for development of the Raydiant fetal pulse oximeter algorithm.

SUMMARY:
The objective of this study is to collect and compare fetal SpO2 waveforms and reference values to inform algorithm development for signal qualification and FSpO2 calculations. Subjects are women in labor.

DETAILED DESCRIPTION:
The Raydiant Data Collection System (DCS) captures red and infrared waveforms that can be post-processed to calculate fetal functional oxygen saturation of arterial oxygen saturation (SpO2) and pulse rate. These waveforms are acquired from the fetus when the sensor is placed at the cheek, temple, or forehead. Acquisition of these waveforms is a necessary step toward signal qualification and data processing algorithms. The Raydiant DCS is a similar device to the original Nellcor N-400 System. Clinical research with the N-400 System demonstrated that fetal pulse oximetry values provide 54.2% positive predicative value and 92.9% sensitivity for detecting newborn metabolic acidosis (defined by pH<7.15).1 This provided a significant aid to clinicians for diagnosing endangering states of fetal hypoxia.

In this study, both the participants and the health-care providers are blinded to the oximetry data; therefore, clinical decisions regarding interventions are made based on routine clinical monitoring. The primary analysis will be performed by comparing the post-processed waveforms. Other than device placement and a period of monitoring not to exceed 6 hours, there is no change to the standard of care procedures for fetal monitoring. As stated above, the sensor displays will not be used to guide or alter patient management.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable of providing informed consent.
2. Age > 18 years.
3. Gestational age > 36 weeks.
4. Singleton pregnancy.
5. Vertex presentation,
6. In latent or active labor,
7. Category I or II tracings,
8. Epidural anesthesia, and
9. Ruptured amniotic sac with cervical dilation of >2 cm and a station of -2 or lower.

Exclusion Criteria:

1. Age < 18 years.
2. Gestational age < 36 weeks
3. Multiple gestation
4. Nonvertex fetal presentation
5. Suspected vasa previa
6. Category III CTG tracing
7. Fetal anomalies and/or chromosomal disorders
8. Chorioamnionitis
9. Placenta previa
10. HIV, genital Herpes, or other infection precluding transvaginal monitoring
11. Unable to provide informed consent (e.g., cognitively impaired)
12. Low anterior placenta, or
13. Any condition (temporary or permanent) in which the investigator deems the patient unsuitable for the study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in labor
Enrollment: 15 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of device-related adverse events | Periprocedural
  Rate of device-related adverse events such as erythema or rash

SECONDARY OUTCOMES:
Maternal Outcomes | Periprocedural
  Maternal adverse outcomes such as chorioamnionitis or endometritis
Neonatal Outcomes | Periprocedural
  Apgar Scores at 1 and 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Perry S Barrilleaux, MD, Principal Investigator — Louisiana State University Health Shreveport
Locations (1):
- LSU Health Science Center-Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is available to Raydiant Oximetry and LSU Study Staff only.